CLINICAL TRIAL: NCT04268992
Title: Effect of Long-term Exercise on Haemostasis and Inflammation Compared With Standard Care in Patients With Stable Coronary Artery Disease: a Randomised Clinical Trial
Brief Title: Effect of Long-term Exercise on Haemostasis and Inflammation in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: National Hospital of the Faroe Islands (Other Government)
Responsible Party: Principal Investigator, Jacobina Kristiansen, M.D., PhD-student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-16-02-408-19
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease; Exercise; Inflammation; Hemostasis
Keywords: Cardiovascular Diseases; Exercise; Hemostasis; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term exercise (Experimental): Supervised exercise training three times a week for three months.
  Interventions: Other: Long-term exercise
- Usual care (No Intervention): Patients are not offered supervised exercise.

INTERVENTIONS:
Other: Long-term exercise — All patients randomised to long-term exercise will perform exercise training at least three times a week for three months. The exercise is supervised and individualised.
  Arms: Long-term exercise

SUMMARY:
Introduction: Regular exercise training improves prognosis in patients with coronary artery disease (CAD). This study investigates whether the beneficial effects of exercise can be partly explained by favourable changes in haemostasis and inflammation.

Methods: 150 CAD patients are randomised to a supervised long-term exercise program (3 months) or usual care. Blood samples are obtained at baseline, 1.5 months, and 3 months after randomisation.

Results: The investigators will evaluate platelet turnover and aggregation, coagulation, fibrinolysis, and inflammatory markers before and after short- and long-term exercise, and the two randomised groups will be compared.

Perspectives: The present study will increase our knowledge of the beneficial mechanisms underlying the effect of exercise in CAD patients, potentially paving the way for improved exercise recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Angiographically verified coronary artery disease with stenosis of at least 50% or previous percutaneous coronary intervention (PCI)/coronary artery bypass graft (CABG) surgery.
* Diagnosis or revascularisation have been made at least 12 months prior to inclusion.

Exclusion Criteria:

* Inability to perform strenuous exercise
* Anticoagulant treatment
* Heart failure (ejection fraction <30% or NYHA >2)
* Implanted implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT)
* Serious arrhythmia requiring hospitalisation within the last 6 months
* Severe valvular heart disease
* Chronic obstructive pulmonary disease GOLD IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Changes in fibrinolytic biomarkers: tissue plasminogen activator (t-PA) and plasminogen activator inhibitor-1 (PAI-1). | 3 months
  Changes in fibrinolytic biomarkers in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare fibrinolytic biomarkers assessed at baseline and after three months of supervised exercise for every patient.
Changes in clot maximum absorbance using the clot lysis assay. | 3 months
  Changes in maximum absorbance in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare clot maximum absorbance assessed at baseline and after three months of supervised exercise for every patient.
Changes in clot lysis time using the clot lysis assay. | 3 months
  Changes in clot lysis time in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare clot lysis time assessed at baseline and after three months of supervised exercise for every patient.
Changes in area under the curve using the clot lysis assay. | 3 months
  Changes in area under the curve in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare area under the curve assessed at baseline and after three months of supervised exercise for every patient.

SECONDARY OUTCOMES:
Changes in platelet aggregation using arachidonic acid (ASPI) as agonist. | 3 months
  Changes in platelet aggregation with ASPI as agonist in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in platelet aggregation using adenosine diphosphate (ADP) as agonist. | 3 months
  Changes in platelet aggregation with ADP as agonist in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in platelet aggregation using thrombin receptor activating peptide-6 (TRAP) as agonist. | 3 months
  Changes in platelet aggregation with TRAP as agonist in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in thrombin generation assessing lag-time until initial thrombin generation. | 3 months
  Changes in lag-time until initial thrombin generation in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in thrombin generation assessing maximum concentration of thrombin. | 3 months
  Changes in maximum concentration of thrombin in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in thrombin generation assessing time to peak. | 3 months
  Changes in time to peak in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in thrombin generation assessing endogenous thrombin potential. | 3 months
  Changes in endogenous thrombin potential in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare the results assessed at baseline and after three months of supervised exercise for every patient.
Changes in coagulation biomarkers: APTT, INR, Factor VIII, vWF. | 3 months
  Changes in coagulation biomarkers in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare coagulation biomarkers assessed at baseline and after three months of supervised exercise for every patient.
Changes in inflammatory biomarkers: CRP, multiple interleukins, tumor necrosis factor alpha (TNF-α), interferon gamma (INF-γ) and more. | 3 months
  Changes in inflammatory biomarkers in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group). Moreover, the investigators will compare inflammatory biomarkers assessed at baseline and after three months of supervised exercise for every patient.

OTHER OUTCOMES:
Changes in cardiorespiratory performance: maximal oxygen uptake | 3 months
  Changes in maximal oxygen uptake in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group).
Changes in cardiorespiratory performance: maximal power output | 3 months
  Changes in maximal power output in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group).
Changes in physical health and mental health (quality of life) assessed by the SF-36v2 questionnaire. | 3 months
  Changes in physical and mental health in coronary artery disease patients who are randomised to long-term exercise compared with patients randomised to usual care (control group).
Incidence of adverse events associated with the exercise intervention. | 3 months
  Number of adverse events (severe, moderate or mild) and training related injuries in coronary artery disease patients who are randomised to long-term exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital of the Faroe Islands, Tórshavn, Faroe Islands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kristiansen J, Kristensen SD, Hvas AM, Ellingsgaard H, Mohr M, Grove EL, Sjuretharson T. Effects of Acute Exercise and 12-Week High-Intensity Interval Training on Inflammatory Biomarkers in Stable Coronary Artery Disease: A Randomized Controlled Trial. J Am Heart Assoc. 2026 Feb 3:e042256. doi: 10.1161/JAHA.125.042256. Online ahead of print. PMID 41631762
- [Derived] Sjuretharson T, Kristiansen J, Nordsborg NB, Gregersen NO, Lydersen LN, Grove EL, Kristensen SD, Hvas AM, Mohr M. The angiotensin-converting enzyme I/D polymorphism does not impact training-induced adaptations in exercise capacity in patients with stable coronary artery disease. Sci Rep. 2023 Oct 25;13(1):18300. doi: 10.1038/s41598-023-45542-0. PMID 37880303
- [Derived] Kristiansen J, Grove EL, Sjuretharson T, Rasmussen J, Mohr M, Kristensen SD, Hvas AM. Haemostasis and fibrinolysis after regular high-intensity interval training in patients with coronary artery disease: a randomised controlled trial. Open Heart. 2022 Nov;9(2):e002127. doi: 10.1136/openhrt-2022-002127. PMID 36428083
- [Derived] Kristiansen J, Sjuretharson T, Grove EL, Rasmussen J, Kristensen SD, Hvas AM, Mohr M. Feasibility and impact of whole-body high-intensity interval training in patients with stable coronary artery disease: a randomised controlled trial. Sci Rep. 2022 Oct 14;12(1):17295. doi: 10.1038/s41598-022-21655-w. PMID 36241898